CLINICAL TRIAL: NCT00003005
Title: A Phase I Study of Cordycepin (NSC 63984) Plus 2'-Deoxycoformycin (NSC 218321) in Patients With Refractory TdT-Positive Leukemia
Brief Title: Chemotherapy With Cordycepin Plus Pentostatin in Treating Patients With Refractory Acute Lymphocytic or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065572; BUMC-4266; NCI-T96-0051
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2000-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; TdT positive adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — cordycepin; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- deoxycoformycin and cordycepin (Experimental): Dose escalation for deoxycoformycin and cordycepin
  Interventions: Drug: Cordycepin; Drug: Deoxycoformycin

INTERVENTIONS:
Drug: Cordycepin — Dose escalation study using the following doses:
  6mg/m2, 12 mg/m2, 24mg/m2, 48mg/m2
Drug: Deoxycoformycin — Dose escalation using the Fibonacci dose escalation sequence starting dose 2mg/m2, escalating to 3mg/m3 intravenous
  Other Names: pentostatin, dCF

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy consisting of cordycepin plus pentostatin in treating patients with refractory acute lymphocytic or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety, maximum tolerated dose, adverse effects, and toxicities of cordycepin, given 1 hour following a fixed dose of the adenosine deaminase inhibitor pentostatin, in patients with refractory TdT positive leukemia. II. Determine the single and multiple dose pharmacokinetics of cordycepin given 1 hour following a fixed dose of pentostatin. III. Characterize selected whole blood and blast cell metabolic parameters serially in relation to cordycepin/pentostatin administration. IV. Measure and quantify any clinical responses in refractory TdT positive leukemia patients following cordycepin/pentostatin administration.

OUTLINE: This is a dose escalation study. Each treatment course is 28 days in length. On days 1-3 pentostatin is administered over 5 minutes by IV bolus and followed 1 hour later by a 1 hour infusion of cordycepin IV. An escalating dose of pentostatin is given with a fixed dose of cordycepin until the desired level of adenosine deaminase inhibition is observed. After this is determined, a dose escalation schedule for cordycepin is initiated to determine the maximum tolerated dose (MTD) when given in combination with pentostatin. The MTD is determined by the number of patients who exhibit dose limiting toxicity and the severity of the toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: TdT positive acute lymphocytic leukemia or blastic chronic myelogenous leukemia Failed at least one standard treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky greater than 70% Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL Transaminases no greater than 2.5 times normal Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance greater than 60 mL/min Cardiovascular: Ejection fraction greater than 40% Other: Not pregnant or nursing No serious concurrent illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since radiation therapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-12; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days
  Dose limiting toxicities will be assessed within the first 28 days of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Ernst, MD, Study Chair — Boston Medical Center
Locations (13):
- United States (13):
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon